CLINICAL TRIAL: NCT02208882
Title: Randomized, Double-Blind, Placebo-Controlled Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Oral Doses of BMS-986120 in Healthy Subjects and the Effect of BMS-986120 on the Pharmacokinetics of Midazolam in Healthy Subjects
Brief Title: Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BMS-986120 in Healthy Subjects and the Effects of Co-Administration of Midazolam and BMS-986120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CV004-006
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — BMS-986120; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel 1: BMS-986120 or Placebo (Experimental): BMS-986120 or Placebo multiple dose by mouth as specified
  Interventions: Drug: BMS-986120; Drug: Placebo
- Panel 2: BMS-986120 or Placebo (Experimental): BMS-986120 or Placebo multiple dose by mouth as specified
  Interventions: Drug: BMS-986120; Drug: Placebo
- Panel 3: BMS-986120 or Placebo + Midazolam (Experimental): BMS-986120 or Placebo (multiple dose) + Midazolam (single dose) by mouth as specified
  Interventions: Drug: BMS-986120; Drug: Placebo; Drug: Midazolam
- Panel 4: BMS-986120 or Placebo (Experimental): BMS-986120 or Placebo multiple dose by mouth as specified
  Interventions: Drug: BMS-986120; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986120
Drug: Placebo
Drug: Midazolam
  Arms: Panel 3: BMS-986120 or Placebo + Midazolam

SUMMARY:
The purpose of this study is to assess the safety, tolerability and effect on Midazolam pharmacokinetics of multiple oral doses of BMS-986120 in healthy subjects.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. Healthy male and female subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
2. Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI=Weight (kg)/[Height(m)]2
3. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and men, ages 18 to 75, inclusive

Exclusion Criteria:

1. Concurrent, or use within 2-weeks of study drug administration, of marketed or investigational, non-steroidal anti-inflammatory compounds (NSAIDS), aspirin or other antiplatelet agents, oral or parenteral anticoagulants
2. Subjects at screening or prior to first dose with the following abnormal laboratory values upon repeat testing are excluded:

   * i) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >upper limit of normal (ULN)
   * ii) Total bilirubin >ULN, thyroid-stimulating hormone (TSH) >1.5 x ULN with T4 within normal limits (Subjects with mild unconjugated hyperbilirubinemia due to Gilbert's syndrome are excluded)
   * iii) CK >3 x ULN (unless exercise related and CK-MB within normal limits)
   * iv) Activated partial thromboplastin (aPTT) or Prothrombin Time (PT)/International Normalized Ratio (INR) >ULN
   * v) Blood urea nitrogen (BUN) or creatinine (Cr) >ULN
3. Hemoglobin or hematocrit or platelet count <lower limit of normal (LLN)
4. Bleeding time exceeding 8 minutes at pre-dose on Day -1
5. Subjects with micro- or macro-hematuria and/or fecal occult blood detected during screening, baseline or documented during other recent medical assessment, unless deemed not clinically significant by the Investigator and Medical Monitor
6. Any significant acute or chronic medical illness
7. Current or recent (within 3 months of study drug administration) gastrointestinal disease
8. Any major surgery within 12 weeks of study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured by number of subjects experience serious adverse events, deaths, adverse events leading to discontinuation, and potential clinically significant changes in electrocardiogram (ECG) parameters | Up to 168 days
Safety and tolerability measured by percent of subjects experience serious adverse events, deaths, adverse events leading to discontinuation, and potential clinically significant changes in electrocardiogram (ECG) parameters | Up to 168 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986120, BMT-141464, Midazolam, and 1'hydroxymidazolam | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Time of maximum observed plasma concentration (Tmax) of BMS-986120, BMT-141464, Midazolam, and 1'hydroxymidazolam | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Area under the concentration-time curve from time zero to 24h [AUC(TAU)] of BMS-986120 and BMT-141464 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Concentration at the end of the dosing Interval (Ctau) of BMS-986120 and BMT-141464 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Half-life (T-HALF) of BMS-986120 and BMT-141464 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Apparent total body clearance (CLT/F) of BMS-986120, Midazolam, and 1'hydroxymidazolam | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
AUC accumulation index (AI_AUC) of BMS-986120 and BMT-141464 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Effective elimination half-life that explains the degree of AUC accumulation observed (T-HALFeff_AUC) of BMS-986120 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Ratio of metabolite AUC(TAU) to parent AUC(TAU), corrected for molecular weight [MR_AUC(TAU)] of BMT-141464 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Ratio of metabolite Cmax to parent Cmax, corrected for molecular weight (MR_Cmax) of BMT-141464 | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] of Midazolam and 1'hydroxymidazolam | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of Midazolam and 1'hydroxymidazolam | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Ratio of metabolite AUC(INF) to parent AUC(INF), corrected for molecular weight [MR_AUC(INF)] of 1'hydroxymidazolam | Part A (Days 1-8), Part B/C (Days 1-19), & Part D (Days 1-22)
Change from baseline in protease-activated receptor-4 - agonist peptide (PAR4-AP) induced platelet aggregation of BMS-986120 | Part A (Days 1-3) & Part B/C (Days 1-19)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- [Derived] Merali S, Wang Z, Frost C, Callejo M, Hedrick M, Hui L, Meadows Shropshire S, Xu K, Bouvier M, DeSouza MM, Yang J. New oral protease-activated receptor 4 antagonist BMS-986120: tolerability, pharmacokinetics, pharmacodynamics, and gene variant effects in humans. Platelets. 2022 Oct 3;33(7):969-978. doi: 10.1080/09537104.2022.2088719. Epub 2022 Jun 26. PMID 35758258
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx